CLINICAL TRIAL: NCT02599727
Title: Effects of Isometric Exercises on Balance, Heart Rate, Pulse Ox and Blood Pressure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistics reason at the data collection site
Sponsor: Carrick Institute for Graduate Studies (Other)
Responsible Party: Principal Investigator, Frederick Carrick, PhD, FACCN, Principal investigator, Carrick Institute for Graduate Studies
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: CI-IRB-20151104002
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Exercise, Isometric
Keywords: balance, postural; postural equilibrium; heart rate; blood pressure; pulse oxygenation; mental speed
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Isometric exercise (Experimental): Subjects performing the isometric exercises intervention
  Interventions: Other: Isometric exercises
- No exercise (Active Comparator): Subjects not performing the isometric exercises intervention
  Interventions: Other: No exercise

INTERVENTIONS:
Other: Isometric exercises — subjects will perform specific isometric exercises for 10-20 minutes, three times a week throughout the enrollment period
  Arms: Active Isometric exercise
Other: No exercise — Subjects will go on with their life without any specific isometric exercise regimen during the enrollment period
  Arms: No exercise

SUMMARY:
Determine the effects repeated isometric exercises have on balance, blood pressure, heart rate and pulse ox. Another outcome measure will be a mental speed test (how quickly a subject can process information and make decisions based upon that information).

DETAILED DESCRIPTION:
Subjects will complete a mental speed test and will undergo Computerized Dynamic Posturography (CDP) testing using the modified Clinical Testing of Sensory Integration in Balance (mCTSIB) protocol: the subjects will be required to stand on a hard or compliant surface (a 4" tall foam cushion of known mechanical properties) in a comfortable posture, feet shoulder width, with eyes open or closed, head straight and arms to the side and free to move, gazing forward, and breathing normally. Immediately prior to the CDP testing, subjects will have their heart rate, blood pressure and pulse Ox measured. These will constitute the baseline information.

Subjects will then be divided into two groups: the isometric exercise group (they will be instructed to perform specific isometric exercises three times a week, for the next 8 weeks) and the control group (no exercises will be prescribe to them).

The same testing procedure indicated above will be followed at the end of the 8 weeks. The mental speed test, CDP testing, heart rate, blood pressure and pulse Ox will constitute the follow-up information.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals

Exclusion Criteria:

* Any pathology preventing the subject to safely perform the isometric exercises (the clinician enrolling the subjects will make the decision)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Changes in Heart Rate | Baseline and at 8 weeks
  Changes in heart rate at rest will be assessed between baseline (at enrollment) and after the treatment period. It will be used to investigate if isometric exercises affect it and how much.

SECONDARY OUTCOMES:
Changes in Stability Score | Baseline and at 8 weeks
  The Stability Score is calculated as percentage ratio of the actual sway and the theoretical limit of stability.
  Changes in Stability Score will be assessed between baseline (at enrollment) and after the treatment period. It will be used to investigate if isometric exercises affect it and how much.
Changes in Blood Pressure | Baseline and at 8 weeks
  Changes in Blood pressure (measured in standard conditions) will be assessed between baseline (at enrollment) and after the treatment period. It will be used to investigate if isometric exercises affect it and how much.
Changes in Mental Speed | Baseline and at 8 weeks
  The subject will be presented a series of word/image pairs and/or simple mathematical equations or number sequences. If a pair matches, the subject has to click the "Correct" button, if the pair does not match, the "Incorrect" button . However, if the word "Opposite" appears at the top of the screen, the asnwer needs to be reversed. The subject has up to 5 minutes to complete the task.
  The Accuracy of the answers expressed as percentage will be used as measure of mental speed. Changes in Accuracy will be assessed between baseline (at enrollment) and after the treatment period. It will be used to investigate if isometric exercises affect it and how much.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick R Carrick, PhD, Principal Investigator — Carrick Institute for Graduate Studies
Locations (1):
- Carrick Institute for Graduate Studies, Cape Canaveral, Florida, United States